CLINICAL TRIAL: NCT01342562
Title: The Effects of Intrathecal Dexmedetomidine on Spinal Anesthesia Using Diluted Low-Dose Bupivacaine for Transurethral Resection of Prostate in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2010-0513
Record Dates: First submitted 2011-04-15; First posted 2011-04-27 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Benign Prostatic Hypertrophy
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DXM-bupivacaine (Experimental)
  Interventions: Drug: spinal anesthesia
- saline-bupivacaine (Placebo Comparator)
  Interventions: Drug: spinal anesthesia

INTERVENTIONS:
Drug: spinal anesthesia — 0.4% bupivacaine(normal saline 0.3ml with dexmedetomidine 3 mcg)
  Arms: DXM-bupivacaine
Drug: spinal anesthesia — 0.4% bupivacaine(normal saline 0.3 ml with 0.5% bupivacaine 1.2 ml)
  Arms: saline-bupivacaine

SUMMARY:
Spinal block is the most common anesthetic technique for transurethral resection of prostatectomy (TURP). Most patients undergoing TURP are elderly and frequently present with cardiopulmonary and endocrine diseases. Low-dose local anesthetic is commonly administer to limit the block level to minimize the hemodynamic changes. However, sometimes it may not provide an adequate level of sensory block. Thus, intrathecal additive is frequently administer with local anesthetic to improve analgesic effect.

Dexmedetomidine(DXM), a selective 2-adrenoreceptor agonist, has been used in the epidural space in humans without any reports of neurological deficits. Previous clinical studies showed that intravenous dexmedetomidine administration prolonged the sensory and motor blocks of bupivacaine spinal analgesia. But clinical studies about the use of intrathecal DXM with local anesthesia in humans are scarce in the literature. Kanazi et al. found that 3μg DXM added to 12 mg spinal bupivacaine produced the significant short onset of sensory and motor block as well as significantly longer duration of sensory and motor block than bupivacaine. And Al-Mustafa et al. reported that intrathecal dexmedetomidine as an adjuvant to 12.5mg bupivacaine in spinal anesthesia has a dose dependant effect on the onset and regression of sensory and motor block.

In our previous study, low-dose diluted bupivacaine 5 mg provided sufficient anesthetic level when opioid was added with local anesthetic. However, opioid-induced side effects, such as pruritus, nausea, or vomiting, could be an obstacle in common use. The aim of this study is to evaluate whether DXM-low-dose bupivacaine spinal anesthesia can provide the effective spinal anesthesia and postoperative analgesia with minimal side effect compare to the local anesthetic only group.

This study was conducted in a randomized, double-blind, controlled fashion. Patients were randomly allocated to DXM group or Saline group. DMT group received hyperbaric bupivacaine 0.5% (1.2 ml) (6 mg) in dextrose 8% solution + DMT 0.3 ml (3 µg)-in total, bupivacaine 0.4% (1.5 ml) intrathecally and Saline group received hyperbaric bupivacaine 0.5% (1.2 ml) (6 mg) in dextrose 8% solution + normal saline 0.3 ml -in total, bupivacaine 0.4% (1.5 ml) intrathecally. After spinal block, the level of sensory block, defined as the dermatomal segment with loss of pain sensation to pin-prick with a 22 G hypodermic needle and cold sensation to alcohol swab was measured every 2 min after intrathecal injection. The investigators recorded the peak sensory block level, time to peak block level from intrathecal injection, blood pressure and heart rate, and analgesic supplementation during operation. The maximum motor block level was assessed according to the modified Bromage scale. During postoperative period, the frequency of analgesic requirement, time to the first analgesic request, and pain scores were evaluated by blind investigator.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* the patient who undergoing elective TURP for benign prostatic hypertrophy under spinal anesthesia

Exclusion Criteria:

* Past history of spine surgery
* infection focus at back
* coagulopathy
* hypersensitivity to local anaesthetics or DMT
* mental disturbance
* neurological disease

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of efficacy of DXM-bupivacaine | The sensory block level at every 2 minutes (up until 14 minutes) after drug injection during spinal anesthesia
  The primary objective is to evaluate the effects of DXM-bupivacaine in spinal block level compare to the saline-bupivacaine (peak sensory block level, time to peak sensory block level reached).

SECONDARY OUTCOMES:
Comparison of the degree of the postoperative analgesic effect | change in VAS(Visual Analog Scale) at 6 hours and 24 hours after surgery
  Secondary objective is the comparison of the degree of the postoperative analgesic effect between the DXM group and the Saline group (visual analog scale at postoperative 6 hours and 24 hours, time to first analgesic request).

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Kanazi GE, Aouad MT, Jabbour-Khoury SI, Al Jazzar MD, Alameddine MM, Al-Yaman R, Bulbul M, Baraka AS. Effect of low-dose dexmedetomidine or clonidine on the characteristics of bupivacaine spinal block. Acta Anaesthesiol Scand. 2006 Feb;50(2):222-7. doi: 10.1111/j.1399-6576.2006.00919.x. PMID 16430546
- [Background] Elcicek K, Tekin M, Kati I. The effects of intravenous dexmedetomidine on spinal hyperbaric ropivacaine anesthesia. J Anesth. 2010 Aug;24(4):544-8. doi: 10.1007/s00540-010-0939-9. Epub 2010 May 14. PMID 20467879
- [Background] Kaya FN, Yavascaoglu B, Turker G, Yildirim A, Gurbet A, Mogol EB, Ozcan B. Intravenous dexmedetomidine, but not midazolam, prolongs bupivacaine spinal anesthesia. Can J Anaesth. 2010 Jan;57(1):39-45. doi: 10.1007/s12630-009-9231-6. Epub 2009 Dec 29. PMID 20039221
- [Derived] Kim JE, Kim NY, Lee HS, Kil HK. Effects of intrathecal dexmedetomidine on low-dose bupivacaine spinal anesthesia in elderly patients undergoing transurethral prostatectomy. Biol Pharm Bull. 2013;36(6):959-65. doi: 10.1248/bpb.b12-01067. PMID 23727917